CLINICAL TRIAL: NCT06692231
Title: Impact of Hospital Pharmacist Intervention on Medication Management in Dialysis Patients After Assessment of Health Literacy Level
Brief Title: Impact of Hospital Pharmacist Intervention on Medication Management in Dialysis Patients
Acronym: IPhaDia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Vichy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHV-2024-10
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Renal Dialysis; Health Literacy Level; Kidney Disease, Chronic
Keywords: clinical pharmacist; end stage renal disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controle Arm (No Intervention): Control arm: will have no specific intervention
- Intervention Arm (Experimental): Intervention arm: Patient will have an interview with a clinical pharmacist to explain the role of each medication. The pharmacist will also explain the best moment to take each medication.
  Interventions: Behavioral: Pharmacist intervention

INTERVENTIONS:
Behavioral: Pharmacist intervention — Patient will have an interview with a clinical pharmacist to explain the role of each medication. The pharmacist will also explain the best moment to take each medication.
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to learn if an intervention of a hospital pharmacist could help, dialysis patients managed his treatment. In a first time, the health literacy level will be assed.

The main questions it aims to answer are:

What is the impact of the clinical pharmacist intervention on the understanding level and management level of his treatment by the patient? Does the intervention of the pharmacist has an effect on the biologicals parameters of the patient? Researchers will compare a group with a pharmacist intervention VS a group without pharmacist intervention for dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* On dialysis (peritoneal dialysis, hemodialysis) for at least 3 months
* Prescription for at least 5 daily medications
* Patient who has not received any pharmaceutical consultation from a hospital pharmacist as part of his or her treatment for chronic renal failure.

Exclusion Criteria:

* Patient does not speak and/or understand French
* Patient's cognitive state does not permit an interview
* Patient not autonomous in managing his or her daily medication (e.g.: patient in nursing home)
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Level of understanding and treatment management | 12 months
  Assessment of level of understanding and management of treatment using a survey based on the questionnaire validated by the French Health Authority (HAS).
  In order to take better account of the diversity of treatments for dialysis patients, we will use an adaptation of this questionnaire describing more precisely the patient's knowledge of treatments related to phosphocalcic metabolism and potassium.
  A score of 7 on this questionnaire means an excellent understanding of the treatment A score of 0 on this questionnaire means the poorest understanding of the treatment

SECONDARY OUTCOMES:
level of health literacy | 12 months
  Literacy will be assessed measured using the French version of the Short Test of Functional Health Literacy in Adults (STOFHLA).
  STOFHLA scale interpretation:
  Score 0-16: Inability to read and interpret healthcare texts Score 17-22: Problem reading and interpreting healthcare texts Score 23-36: Can read and interpret most healthcare texts
Assessment of patient-reported compliance with medication | 12 months
  The patient-reported compliance will be assed using the GIRERD questionnaire. This tool is made of 6 questions. A score of 0 mean a good compliance and a score ≥3 mean a bad compliance
Kalemia evolution | 12 months
  concentration of potassium in blood plasma
Phosphatemia evolution | 12 months
  concentration of phosphate in blood plasma
Calcemia evolution | 12 months
  concentration of calcium in blood plasma
PTH evolution | 12 months
  concentration of PTH in blood plasma
Vitamine D evolution | 12 months
  concentration of vitamine D in blood plasma
Quality of life | 12 months
  Patients' quality of life will be assessed using the EQ-5D-5L tool. The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each dimension is describe by a five levels scale. (From 0 the worst outcome to 5 the best outcome). A visual analogue scale, where the patient rate is health form 0 to 100, complete this descriptive system.
Assessment of compliance with medication | 12 months
  Call to the patient's usual pharmacy to check that medication retrieval is regular and get the pharmacist's opinion of the patient, by asking the following question: "Based on the last 6 months in your pharmacy's patient file, how would you rate the regularity of this patient's medication retrieval? "Good - Intermediate - Poor".

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier de Vichy, Vichy, France, France

IPD SHARING:
Plan to Share IPD: Undecided